CLINICAL TRIAL: NCT03773094
Title: Effect of Guava Leaves Extract Mouth Wash on Antibacterial Activity, Salivary pH and Patient Satisfaction Compared to Chlorhexidine Mouth Wash in High Caries Risk Patients: A Randomized Control Clinical Trial
Brief Title: Antibacterial Effect of Guava Leaves Extract Mouthwash Compared to Chlorhexidine Mouthwash in High Caries Risk Patients
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Engy Mostafa Magdy Abdou Ahmed Kassem, Assistant Lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Guava leaves extract CHX
Record Dates: First submitted 2018-12-08; First posted 2018-12-12 (Actual); Last update posted 2018-12-12 (Actual); Status verified 2018-12

CONDITIONS: High Caries Risk Patients; Antimicrobial Effect; Salivary pH; Patient Satisfaction to Taste
MeSH Terms: interventions — Chlorhexidine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Guava leaves extract (Experimental): A natural product that is prepared as a mouthwash
  Interventions: Drug: Guava leaves extract
- Chlorhexidine (Active Comparator): chemical agent Chlorhexidine as a mouthwash
  Interventions: Drug: Chlorhexidine

INTERVENTIONS:
Drug: Guava leaves extract — Natural product : The leaves of the guava tree are full of antioxidants, anti-inflammatory agents, antibacterials, and even tannins that can have significant health benefits, from treating stomach troubles to chronic diseases like cancer
  •
  Other Names: Psidium guajava
  Arms: Guava leaves extract
Drug: Chlorhexidine — chemical agent used as a mouthwash against cariogenic bacteria. considered the gold standard
  Other Names: Chlorhexidine glucnate
  Arms: Chlorhexidine

SUMMARY:
This trial is to test the antibacterial effect of Guava leaves extract mouth wash compared to Chlorhexidine mouth wash in high caries risk patients.

Also salivary pH and patient satisfaction to taste will also be tested.

DETAILED DESCRIPTION:
This study is conducted to evaluate the effect of Guava leaves extract mouth wash on anti-bacterial activity against streptococcus mutans, salivary pH and patient satisfaction to taste compared to Chlorhexidine mouth wash.

P: Population with high caries risk patients I: Intervention by Guava leaves extract mouthwash C: Control is Chlorhexidine mouthwash O1: The primary outcome is antibacterial activity. O2: The secondary outcome is salivary pH O3: The tertiary outcome is patient satisfaction to taste

ELIGIBILITY:
Inclusion Criteria

1. High caries risk patients
2. 18-50 years
3. Healthy cooperative patients
4. Males or Females

Exclusion Criteria

1. Medically compromised patients
2. Patients with any systemic disease that might affect the salivary flow
3. Allergy to any of the ingredients
4. Patients with physical limitations that might affect normal tooth brushing and mouth rinsing
5. Presence of intraoral infections
6. Currently using any mouth rinse
7. Smokers
8. Use of antibiotics in the previous 30 days

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 94 (Estimated)
Dates: Start 2019-01 (Estimated); Primary Completion 2019-11 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
Anti-bacterial effect against streptococcus mutans | 3 months
  Antimicrobial effect against streptococcus mutans: saliva samples collected and total bacterial count measured after agar plates incubating, expressed in colony forming units

SECONDARY OUTCOMES:
Salivary pH | 3 months
  Saliva samples pH will be measured using digital pH meter to evaluate its efficacy in preventing the action of acidogenic bacteria in high caries risk patients.
  It displays numerical value.

OTHER OUTCOMES:
Patient satisfaction to taste: questionnaire | 3 months
  The patient will fill a questionnaire to assess patient satisfaction to taste after usage of the mouthwash. Nominal answers

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gupta D, Nayan S, Tippanawar HK, Patil GI, Jain A, Momin RK, Gupta RK. Are herbal mouthwash efficacious over chlorhexidine on the dental plaque? Pharmacognosy Res. 2015 Jul-Sep;7(3):277-81. doi: 10.4103/0974-8490.155874. PMID 26130940
- [Background] Ravi K, Divyashree P. Psidium guajava: A review on its potential as an adjunct in treating periodontal disease. Pharmacogn Rev. 2014 Jul;8(16):96-100. doi: 10.4103/0973-7847.134233. PMID 25125881
- [Background] Singla S, Malhotra R, Nd S, Saxena S. Antibacterial Efficacy of Mouthwash Prepared from Pomegranate, Grape Seed and Guava Extracts against Oral Streptococci: An in Vivo Study. J Clin Pediatr Dent. 2018;42(2):109-113. doi: 10.17796/1053-4628-42.2.5. Epub 2017 Oct 31. PMID 29087796
- [Background] Shah S, Bargale S, Dave BH, Deshpande A, Kariya PB, Karri A. Comparison of Antimicrobial Efficacy of (between) 0.2% Chlorhexidine and Herbal Mouthwash on Salivary Streptococcus mutans: A Randomized Controlled Pilot Study. Contemp Clin Dent. 2018 Jul-Sep;9(3):440-445. doi: 10.4103/ccd.ccd_264_18. PMID 30166841
- [Background] Jain I, Jain P. Comparative evaluation of antimicrobial efficacy of three different formulations of mouth rinses with multi-herbal mouth rinse. J Indian Soc Pedod Prev Dent. 2016 Oct-Dec;34(4):315-23. doi: 10.4103/0970-4388.191409. PMID 27681394